CLINICAL TRIAL: NCT07132840
Title: Immediate Effects of Balance Training Combined With Kinesio-taping on Static Balance, Dynamic Balance and Proprioception in People With Functional Ankle Instability (FAI)- A Quasi-experimental Study
Brief Title: Combined Effects of Balance Training and Taping in People With Functional Ankle Instability.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. John's Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TH-41/2023
Record Dates: First submitted 2025-08-13; First posted 2025-08-20 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Chronic Ankle Instability; Functional Ankle Instability; Lateral Ankle Sprain
Keywords: lateral ankle sprain; functional ankle instability; kinesiotape; balance training; proprioception; balance error scoring system; star excursion balance test; cumberland ankle instability tool; joint position sense

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group- Balance training combined with kinesio tape (Experimental): Participants with functional ankle instability received balance training on various unstable surfaces after kinesio tape application.
  Interventions: Procedure: Kinesio tape application followed by single session of balance training on various unstable surfaces.

INTERVENTIONS:
Procedure: Kinesio tape application followed by single session of balance training on various unstable surfaces. — Participants with functional ankle instability received balance training on various unstable surfaces after kinesio tape application.

SUMMARY:
Approximately 70% of all people who have had a simple ankle sprain tend to develop continuing instability and pain. Chronic ankle instability is the most common problem that impairs the patients' daily functions. This can lead to balance issues, chances of recurrent sprain and loss of function.

* Therefore, the investigators are conducting this study to assess the immediate effects of balance exercises along with kinesio-taping on static balance, dynamic balance and joint position sense, and to also assess if this combination can be used as stopgap (quick-fix) to improve balance and proprioception before a session of sports activity in people involved in recreational sports.
* During the study, the participants will receive a one-time application of ankle kinesio-taping followed by an hour of balance training exercises on different surfaces such as Dynair, Bosu, Foam pads, and Mini tramp. Joint position sense will be assessed using a digital inclinometer that is already available in the department.
* The participants will be tested using certain physical tests to assess the static balance and dynamic balance using the Balance Error Scoring System tool and Star Excursion Balance Test respectively which they will perform before and 24 hours post training.

DETAILED DESCRIPTION:
Ankle sprains account for approximately 85% of lower extremity injuries. Ankle sprains are often incorrectly considered to be harmless injuries with no lasting consequences, but in fact, reduced physical activity, patient reported disability, increased symptoms and risk of re-injury and recurrent injury are all commonly reported months and sometimes even years after the first sprain. Close to 70% of those who have suffered an ankle sprain develop ankle instability or "giving way" of the ankle during functional activities . There is also evidence suggesting that repetitive ankle sprains are a risk factor for ankle osteoarthritis. The initial injury may result in 2 types of dysfunctions, mechanical instability or functional instability, this influences the outcome by resulting in either i) recovery from the acute sprain or ii) development of chronic instability.

Functional Ankle Instability [FAI], refers to the sensorimotor and neurological deficits that accompany ligamentous injury. Functional Ankle Instability is used to describe the feeling of their ankle giving way, being more painful and being weaker specifically while performing some activity, compared to before the injury. Functional Ankle Instability has been difficult to measure reliably, until recently. Cumberland Ankle Instability Tool is a 9-item 30-point scale developed specifically to measure the severity of Functional Ankle Instability. The CAIT tool has an 83% sensitivity and 75% specificity . In the acute stage, use of the RICE (Rest, Ice, Compression, and Elevation) protocol is recommended to decrease edema, followed by electro modalities such as electrostimulation, ultrasonic therapy, massage, and manual therapy to decrease pain and speed functional recovery .

The essence of evidence-based practice lies in the effectiveness of the treatment that is being provided. Balance training is one such practice currently being used in patients with Functional Ankle Instability [3]. Balance training has been hypothesized to work by activating the mechanoreceptors present in the joint capsule and ligaments of the ankle, which in turn increases the sensory output . These Balance exercises are also found to improve proprioception and thereby improve performance and a sense of stability in individuals with FAI. In addition to these exercises, various external supports are available that help reduce the instability, such as Kinesiotape, brace and much more. Kinesiotape is a cotton strip that is compatible with the skin and is able to stretch up-to 140% its original length. It is a low cost, conveniently accessible tool that can be used to treat various conditions as well as facilitate muscle activity, provide joint stability, postural control and improve physical performance .

Some of the authors have suggested that KT works because of its ability to increase the number of motor units recruited in the muscle. The skin folds due to the increased nature of its elasticity, resulting in increased space below the skin improving circulation and lymphatic drainage. KT has shown improvement in static balance as measured using Balance Error Scoring System . However, there is contradicting and highly inconsistent literature on the effectiveness of KT in improving proprioception, balance Range of Motion in people with Functional ankle instability .

There have been some studies that have focused on the effects of KT and balance exercises on postural control and balance in athletic population . Most of these studies have focused on athletes in organized sports, leaving out the remainder of the population, majority of whom are recreational players. Consequently, there is a need for more research in this population as these are the people who most often do not undergo any type of sports specific training or get any type of rehabilitation post-injury. These are the people who ignore their injuries and its symptoms simply because they do not have the time or sometimes, the money to avail proper rehabilitation due to their hectic work life.

Therefore, this study focuses on the immediate effects of KT combined with balance training on balance and proprioception in the non-athletic, recreational sports population. This following study is also being conducted to see if the combination of KT and Balance training can be used as a stopgap treatment strategy before a session of recreational sport activity.

ELIGIBILITY:
Inclusion Criteria:

* Adults between the age of 18 - 40 years with a history of at least 1 ankle sprain
* Cumberland Ankle Instability Test score of ≤ 27 indicative of Functional Ankle instability
* No episode of an ankle sprain in the past 3 months
* No history of limb fracture in the past 6 months prior to study
* Absence of vestibular disorders or concussion symptoms
* No history of any neuromuscular disorders

Exclusion Criteria:

* Health issue that would interfere with participants safety during exercise
* Participants with active malignancy, cellulitis, skin infection, or open wound.
* Presence of common cold.
* After Inclusion in study:

  * Participants excluded if they missed the 24 hours follow up.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-09-21 (Actual); Primary Completion 2024-01-25 (Actual); Study Completion 2024-01-25 (Actual)

PRIMARY OUTCOMES:
Balance error scoring system (BESS)- for static balance | 24 hours from the recruitment
Star excursion balance test (SEBT)- for dynamic balance | 24 hours from recruitment

SECONDARY OUTCOMES:
Active joint position reproduction test using digital inclinometer- for proprioception | 24 hours from recruitment

CONTACTS AND LOCATIONS:
Locations (1):
- St. John's Medical college & Hospital, Bangalore, Karnataka, India

IPD SHARING:
Plan to Share IPD: Undecided